CLINICAL TRIAL: NCT02332109
Title: ODM 5 in the Treatment of Corneal Edematous Fuchs' Endothelial Dystrophy
Status: Completed | Type: Observational
Sponsor: TRB Chemedica AG (Industry)
Responsible Party: Sponsor
Other Study IDs: ODM5FDE-PMCF-DE-2015-01
Record Dates: First submitted 2014-12-19; First posted 2015-01-06 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Fuchs' Endothelial Dystrophy; Corneal Edema
Keywords: Fuchs endothelial dystrophy; oedema; sodium chloride; hyaluronan; sodium hyaluronate
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy; Corneal Edema; Edema

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ODM 5-group
  Interventions: Device: ODM 5

INTERVENTIONS:
Device: ODM 5 — ODM 5 is a CE-certified, preservative-free, hyperosmolar ophthalmological solution containing 5% sodium chloride and 0.15% sodium hyaluronate recommended for the reduction of corneal edema. The patient will use ODM 5 on a daily basis in accordance with the instructions for use and as recommended by the investigator over a period of 8 weeks.

SUMMARY:
Clinical observation to confirm the clinical safety and efficacy of ODM 5 in the treatment of corneal edema caused by Fuchs' endothelial dystrophy.

DETAILED DESCRIPTION:
Patients with a Fuchs' endothelial dystrophy-induced corneal edema and an ODM 5 therapy recommendation prior to their inclusion will be observed in normal practice setting in this post-market clinical follow-up study. In this indication, the use of ODM 5 should extract the fluid excess in the cornea away by an osmotic effect, enabling the cornea to temporarily regain a normal state of hydration. As a consequence, the patient's visual acuity, contrast perception, corneal thickness and ocular complaints/symptoms should improve. The hyaluronan in ODM 5 helps to protect and heal the cornea in case of irritation and thus, enables the cornea to regain a normal state of hydration and participates in improving the quality of vision.

ELIGIBILITY:
Inclusion Criteria:

* Presence of corneal oedema caused by Fuchs' endothelial dystrophy
* Existing ODM 5 recommendation prior to inclusion

Exclusion Criteria:

* Contact lens wear
* Hypersensitivity to one of the ODM 5 components
* Appointment for eye surgery within 8 weeks after date of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a Fuchs endothelial dystrophy-induced corneal edema and an ODM 5 therapy recommendation.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2015-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Visual acuity (both eyes) | Day 56
  Measurement of uncorrected and best corrected visual acuity (both eyes)

SECONDARY OUTCOMES:
Corneal thickness | Day 0, day 28 and day 56
  Measurement of central corneal thickness (both eyes)
Visual acuity (both eyes) | Day 0 and day 28
  Measurement of uncorrected and best corrected visual acuity (both eyes)
Contrast perception (Measurement of contrast values (both eyes)) | Day 0, day 28 and day 56
  Measurement of contrast values (both eyes)
Subjective ocular complaints and symptoms (11-point Likert scale) | Day 0, day 28 and day 56
  The following ocular complaints or symptoms will be evaluated on an 11-point Likert scale ranging from '0' (no complaints) to '10' (maximum complaints):
  * glare sensitivity
  * burning
  * foreign body sensation
  * halos
  * pruritus
  * blurred vision
  * redness
  * pain
  * tingling
  * stitching
  * dryness
  * watering eyes
Safety parameter (Adverse events) | Day 0, day 28 and day 56
  Adverse events judged to be unexpected and (possibly) related to ODM 5 will be documented

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (4):
  - Universitätsklinikum Düsseldorf, Augenklinik, Düsseldorf
  - Praxis Dr. Thomas Kaercher, Heidelberg
  - Universitätsklinikum Magdeburg A.ö.R., Universitätsaugenklinik, Magdeburg
  - Augenklinik der Ludwig-Maximilians-Universität (LMU), Klinikum der Universität München, München